CLINICAL TRIAL: NCT03567551
Title: Novel Biomarkers of Preeclampsia: Aquaporin, Fatty Acid, and S100B
Brief Title: Novel Biomarkers of Preeclampsia, Aquaporin, Fatty Acid, and S110B
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Tekuila Carter, Principal Investigator, University of Alabama at Birmingham
Other Study IDs: IRB-160822006
Record Dates: First submitted 2018-05-21; First posted 2018-06-26 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Pregnancy; Complications; Eclampsia; Aquaporin; Aquaporin 4
MeSH Terms: conditions — Pre-Eclampsia; Eclampsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women w/ Preeclampsia w/o Visual Disturbances or Headache: Preeclampsia Without either Visual Disturbances or Headaches Blood Pressure: >Systolic 160 or Diastolic 110
  Interventions: Other: Women w/ Preeclampsia w/o Visual Disturbances or Headache
- Women w/ Preeclampsia w/ Visual Disturbances or Headaches: Preeclampsia With either Visual Disturbances or Headaches Blood Pressure: >Systolic 160 or Diastolic 110
  Interventions: Other: Women w/ Preeclampsia w/ Visual Disturbances or Headaches
- Women w/o Preeclampsia: Normal Pregnancy Blood Pressure: <140/90
  Interventions: Other: Women w/o Preeclampsia

INTERVENTIONS:
Other: Women w/ Preeclampsia w/o Visual Disturbances or Headache — Up to three maternal blood samples collected from each participant, cerebrospinal fluid collected from each participant during spinal or combined spinal/epidural anesthesia, one umbilical cord blood sample obtained from each participant, four placenta samples obtained from each placenta from each participant
  Groups: Women w/ Preeclampsia w/o Visual Disturbances or Headache
Other: Women w/ Preeclampsia w/ Visual Disturbances or Headaches — Up to three maternal blood samples collected from each participant, cerebrospinal fluid collected from each participant during spinal or combined spinal/epidural anesthesia, one umbilical cord blood sample obtained from each participant, four placenta samples obtained from each placenta from each participant
  Groups: Women w/ Preeclampsia w/ Visual Disturbances or Headaches
Other: Women w/o Preeclampsia — Up to three maternal blood samples collected from each participant, cerebrospinal fluid collected from each participant during spinal or combined spinal/epidural anesthesia, one umbilical cord blood sample obtained from each participant, four placenta samples obtained from each placenta from each participant
  Groups: Women w/o Preeclampsia

SUMMARY:
This is a research study designed to help identify preeclampsia in pregnant women earlier, and possibly lead to better treatment for women preeclampsia.

DETAILED DESCRIPTION:
There is a paucity of biomarkers to predict preeclampsia and for predicting the severity of preeclampsia. This study was designed to identify novel biomarkers for both the prediction of preeclampsia in previously normal pregnancies and for the prediction of the severity of preeclampsia in preeclamptic women. The investigators plan to perform targeted testing for markers that the investigators predict based on their findings or based on available published evidence and the investigators also plan testing for novel markers using various approaches such as proteomics, lipidomics and genomics. The targeted markers will include Aquaporin 4 (AQP4), soluble aquaporin fragments, chemokines, and halogenated fatty acids in the plasma and/or spinal fluid. Aquaporin fragments and AQP4 have been hypothesized to correlate with severe headaches which are complications of severe preeclampsia. The investigators found in their murine studies that there is a correlation between the presence of halogenated fatty acids in the plasma and elevated blood pressure in a murine model of preeclampsia. The approaches will complement the targeted analyses to identify novel markers that have not been predicted yet.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 20 years of age
* Greater than 24 weeks of gestation
* Obstetrics/Anesthesia Team had decided that Combined Spinal/Epidural (CSE) or Spinal Anesthesia will be performed

Exclusion Criteria:

* Pre-pregnancy comorbidities:
* hypertension, diabetes, or pulmonary hypertension
* use of steroids, beta blockers, Ca channel antagonist, anticoagulants
* cardiac or vascular conditions
* severe headaches or visual disturbances
* Inability to receive CSE or Spinal Anesthesia
* Chorioamnionitis, fever, bronchitis, pneumonia

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women older than 20 years of age, who meet all inclusion criteria and none of the exclusion criteria, and who are willing and able to sign informed consent documentation, as well as receive a combined spinal/epidural, or a spinal anesthesia regimen.
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-01-13 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Aquaporin 4 protein fragments in maternal blood plasma | Between hospital admission and prior to epidural or combined spinal/epidural anesthesia
  The investigators plan to perform targeted testing for markers that the investigators predict based on their findings or based on available published evidence
S100B protein fragments in maternal blood plasma | Between hospital admission and prior to epidural or combined spinal/epidural anesthesia
  The investigators plan to perform targeted testing for markers that The investigators predict based on their findings or based on available published evidence
Aquaporin 4 protein fragments in cerebrospinal fluid | At the time of spinal or combined spinal/epidural anesthesia
  The investigators plan to perform targeted testing for markers that the investigators predict based on their findings or based on available published evidence
S100B protein fragments in cerebrospinal fluid | At the time of spinal or combined spinal/epidural anesthesia
  The investigators plan to perform targeted testing for markers that the investigators predict based on their findings or based on available published evidence
Aquaporin 4 protein fragments in cord blood and placental samples | Between delivery and 2 hours after delivery
  The investigators plan to perform targeted testing for markers that the investigators predict based on their findings or based on available published evidence
S100B protein fragments in cord blood and placental samples | Between delivery and 2 hours after delivery
  The investigators plan to perform targeted testing for markers that the investigators predict based on their findings or based on available published evidence

SECONDARY OUTCOMES:
Fatty acids in maternal blood | Between hospital admission and prior to epidural or combined spinal/epidural anesthesia
  The investigators plan to perform targeted testing for markers that the investigators predict based on their findings or based on available published evidence
Fatty acids in cord blood and placental samples | Between immediately post-delivery and 2 hours after delivery
  The investigators plan to perform targeted testing for markers that The investigators predict based on their findings or based on available published evidence
Fatty Acids in cerebrospinal fluid | during epidural or combined spinal/epidural anesthesia
  The investigators plan to perform targeted testing for markers that The investigators predict based on their findings or based on available published evidence

CONTACTS AND LOCATIONS:
Overall Officials: Tekuila Carter, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States